CLINICAL TRIAL: NCT03212898
Title: The Influence of Pharmacist Interventions on the Effectiveness of Warfarin Treatment in Elderly Patients From Rural Areas
Brief Title: Pharmacist Interventions in Rural Elderly Warfarin Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slaven Falamić (Other)
Responsible Party: Sponsor-Investigator, Slaven Falamić, Slaven Falamić,MPharm, Prinicipal-Investigator, Slaven Falamić
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SFalamic
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation; Thrombosis; Cardiac Failure; Hemorrhage
Keywords: pharmacist interventions, warfarin, elderly rural patients
MeSH Terms: conditions — Atrial Fibrillation; Thrombosis; Heart Failure; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Specific pharmacist-led anticoagulation care
  Interventions: Other: anticoagulation care
- Control (No Intervention): The control group will receive usual care; no interventions will be administered.

INTERVENTIONS:
Other: anticoagulation care — Patients in the intervention group will: 1) have a repeated pharmacist-led education on all aspects of warfarin treatment; 2) receive enhanced medication instructions and a care and follow up plan; 3) receive a pill box 4) be refered to the GP with proposal for dose change when outside the therapeutic range or therapy modification to avoid drug interactions with warfarin
  Arms: Intervention

SUMMARY:
The primary study goal is to explore the influence of pharmacist interventions on the effectiveness of warfarin treatment in a specific subpopulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Living site of participant outside the city eg. rural site
* Expected duration of warfarin therapy at least 6 months from the inclusion in the study and 3 months before

Exclusion Criteria:

* Hospitalization
* Vegetarianism
* Patients not able to provide an informed consent
* The use of drug that has an X level of clinical significance of interaction with warfarin according to Lexicomp interact base

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range (TTR) | 6 months
  Time in therapeutic range by Rosendaal method (percentage of time in therapeutic range)

SECONDARY OUTCOMES:
Adverse drug reactions | 6 months
  To measure the difference in number and types of adverse drug reactions between the intervention and the control group
Time to adverse drug reaction | 6 months
  To measure the difference in time to adverse drug reactions between the intervention and the control group
International randomised ratio | 6 months
  To measure the difference in patterns of the International randomised ratio between the intervention and the control group
Adherence | 6 months
  To measure the difference in adherence between the intervention and the control group
Quality of life | 6 months
  To measure the difference of the quality of life in the intervention and the control group at the beginning and the end of the study (validated Croatian version of DUKE - Duke anticoagulation satisfaction scale questionaire)
Incidence and influence of clinically significant drug interactions | 6 months
  To measure the incidence of clinically significant drug interactions (defined by the Lexicomp-interact base as degree C and D of clinical significance) and influence of drug interactions on the effectiveness and safety of treatment between the intervention and the control group
Dietary intake of vitamin K | 6 months
  Changes of dietary intake of vitamin K
Acceptance of pharmacist's intervention by the general practitioners | 6 months
  To measure the rate of acceptance of pharmacist's interventions by the general practitioners

CONTACTS AND LOCATIONS:
Overall Officials: Slaven Falamić, MPharm, Principal Investigator — Pharmacy Branka Marušić

REFERENCES:
- [Derived] Falamic S, Lucijanic M, Ortner-Hadziabdic M, Marusic S, Bacic-Vrca V. Pharmacists' interventions improve health-related quality of life of rural older person on warfarin: a randomized controlled trial. Sci Rep. 2021 Nov 9;11(1):21897. doi: 10.1038/s41598-021-01394-0. PMID 34754004